CLINICAL TRIAL: NCT02880514
Title: A Clinical Evaluation of Propel Mini Sinus Implant Placement in the Frontal Sinus Ostia Following In-office Dilation
Brief Title: In-office Placement of the Propel Mini Sinus Implant in the Frontal Sinus Ostia
Acronym: FRONTIER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intersect ENT (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P500-0616
Record Dates: First submitted 2016-08-18; First posted 2016-08-26 (Estimated); Results first posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-11

CONDITIONS: Chronic Sinusitis
Keywords: Frontal Sinus; Balloon Dilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PROPEL Mini Sinus Implant (Experimental): Placement of the Propel Mini Sinus Implant in one frontal sinus ostia (FSO) assigned to the treatment group following in-office balloon dilation
  Interventions: Device: PROPEL Mini Sinus Implant; Procedure: Balloon Sinus Dilation Alone
- Balloon Sinus Dilation Alone (Active Comparator): In-office balloon dilation of the contralateral frontal sinus ostia (FSO) without implant placement
  Interventions: Procedure: Balloon Sinus Dilation Alone

INTERVENTIONS:
Device: PROPEL Mini Sinus Implant — Sinus implant with 370 mcg of mometasone furoate released over 30 days
  Other Names: PROPEL Mini
  Arms: PROPEL Mini Sinus Implant
Procedure: Balloon Sinus Dilation Alone

SUMMARY:
A randomized controlled trial

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blind, intra-patient controlled, multicenter trial with 50 subjects enrolled at up to 15 sites across the United States. Study subjects undergo implant placement on one side following in-office balloon dilation, while the contralateral side undergoes balloon dilation only and serves as a control.

ELIGIBILITY:
Inclusion Criteria

* Patient has provided written informed consent using a form approved by the reviewing IRB.
* Patient is 18 years of age or older.
* Patient is willing and able to comply with protocol requirements.
* Patient has CRS defined as sinonasal inflammation persisting for more than 12 weeks and complains of at least 2 of the 4 following symptoms: nasal blockage/obstruction/congestion, nasal blockage/obstruction/congestion, nasal discharge (anterior/posterior), facial pain/pressure, reduction/loss of smell
* CRS diagnosis confirmed by CT scan within 3 months prior to enrollment
* Bilateral frontal sinusitis confirmed by Lund-Mackay score of ≥1 on each side
* Post-endoscopic sinus surgery, patient has bilateral obstruction of the frontal sinus ostia by scarring and/or polypoid edema.
* Patient is a candidate for an in-office balloon dilation procedure.
* In the opinion of the investigator, treatment with the Propel Mini Sinus Implant as an adjunct to balloon sinus dilation is technically feasible and clinically indicated in the frontal sinus ostia.

Exclusion Criteria:

* Expanded amount of ethmoid sinonasal polyps extending beyond the middle meatus of grade 3 or 4 unless reduced prior to randomization in the study.
* Oral-steroid dependent condition such as chronic obstructive pulmonary disease (COPD) or other conditions.
* Known history of allergy or intolerance to corticosteroids or mometasone furoate.
* Clinical evidence of acute bacterial sinusitis or invasive fungal sinusitis.
* Active viral illness (e.g., flu, shingles).
* Clinical evidence of disease or condition expected to compromise survival or ability to complete follow-up assessments through Day 180 post-procedure.
* Currently participating in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Silvers, Principal Investigator — Madison ENT
Locations (9):
- United States (9):
  - Sacramento ENT, Sacramento, California
  - ENT Assoicates of South Florida, Boca Raton, Florida
  - ENT of Georgia, Atlanta, Georgia
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Associated Surgical Specialists, Covington, Louisiana
  - St. Luke's ENT Specialists, Kansas City, Missouri
  - BreatheAmerica of Albuquerque, Albuquerque, New Mexico
  - Madison ENT, New York, New York
  - Ohio Sinus Institute, Dublin, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 50 participants were recruited across 12 clinical sites.
Pre-assignment Details: An intra-patient control design was employed where left and right frontal sinuses of each patient were randomized to the treatment or control group after successful completion of in-office balloon dilation.
Units Other Than Participants: sinus sides
Groups:
- PROPEL Mini Sinus Implant: Placement of the Propel Mini Sinus Implant in one frontal sinus ostia (FSO) after a successful in-office balloon dilation
- Balloon Sinus Dilation Alone: Successful in-office balloon dilation of the frontal sinus ostia (FSO) without implant placement
Period: Overall Study
Arm/Group | PROPEL Mini Sinus Implant | Balloon Sinus Dilation Alone
Started | 50; 50 sinus sides (A total of 50 subjects with one sinus side assigned to the treatment group) | 50; 50 sinus sides (A total of 50 subjects with one sinus side assigned to the control group)
Completed | 50; 50 sinus sides | 50; 50 sinus sides
Not Completed | 0; 0 sinus sides | 0; 0 sinus sides

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: This study used an intra-patient design with each participant having one sinus side randomized to the treatment group and the other to the control group.
Arm/Group | All Study Participants
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (13.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 49
  Race: Hispanic | 0
  Race: Other | 1
  Race: Black or African American | 0
  Race: American Indian or Alaska Native | 0
  Race: Asian | 0
  Race: Native Hawaiian or other Pacific Islander | 0
Lund-Mackay Total Score [Mean (Standard Deviation); unit: units on a scale] — The Lund-Mackay score is a method of radiologic staging of chronic rhinosinusitis based on computed tomography (CT) where each sinus is assigned a score of 0 (no abnormality), 1 (partial opacification), or 2 (complete opacification). The overall total score is the sum of scores from 6 sinuses on each side and ranges from 0 to 24 with higher score indicating greater disease burden.
  units on a scale | 10.8 (3.67)
Lund-MacKay Frontal Score [Mean (Standard Deviation); unit: units on a scale] — The Lund-Mackay Frontal score is determined based on computed tomography (CT) of the frontal sinus on a 0 to 2 scale where 0 = no abnormality, 1 = partial opacification, and 2 = complete opacification. The frontal score is the sum of scores on the left and right side and ranges from 0 to 4 with higher score indicating greater disease burden.
  units on a scale | 1.2 (0.40)

OUTCOME MEASURES:

1. Primary Outcome: Patency Rate
Description: Patency of the frontal recess/frontal sinus ostia (FSO) was evaluated on a 3-point grading scale from 0 to 2, with 0=Patent, 1=Restenosed/partially occluded, and 2=Occluded. The percentage of sinuses with patency grade 0 and 1 was used to calculate the patency rate.
Time Frame: Day 30
Population: Outcome analyzed using the intent-to-treat population, which consisted of all randomized subjects and sinuses. Patency grade for 10 sinuses (6 treatment, 4 control) were missing as clinical investigators were unable to view the frontal recess/FSO, reducing the number of evaluable subjects to 44 in the treatment group and 46 in the control group.
Measure: Count of Units; unit: sinus sides
Units Other Than Participants: sinus sides
Groups:
- PROPEL Mini Sinus Implant: Placement of the Propel Mini Sinus Implant in the frontal sinus ostia (FSO) after a successful in-office balloon dilation
- Balloon Sinus Dilation Alone: Successful in-office bilateral balloon dilation of the frontal sinus ostia (FSO) without implant placement
Arm/Group | PROPEL Mini Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 44 | 46
Number analyzed (sinus sides) | 44 | 46
sinus sides | 38 | 33
Statistical Analysis 1: Comparison: PROPEL Mini Sinus Implant vs Balloon Sinus Dilation Alone; Test type: Superiority; p = 0.0391, McNemar — P-value not adjusted for multiplicity; McNemar's exact binomial test was employed to obtain the two-sided p-value at alpha level of 0.05

2. Secondary Outcome: Inflammation Score
Description: Inflammation visual analog scale (VAS) from 0 (no visible inflammation) to 100 (severe inflammation, involving significant and extensive erythema and edema and/or hypertrophy and/or polypoid changes)
Time Frame: Day 30
Population: Inflammation score for 7 sinuses (4 treatment, 3 control) were missing as clinical investigators were unable to view the frontal recess/FSO for 3 treatment and 2 control sinuses, and 1 participant with 1 treatment and 1 control sinuses was lost to follow-up.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Sinuses
Groups:
- PROPEL Mini Sinus Implant: Placement of Propel Mini Sinus Implant after a successful in-office balloon dilation of the frontal sinus ostia (FSO)
- Balloon Sinus Dilation Alone: Successful in-office bilateral balloon dilation of the frontal sinus ostia (FSO) only without implant placement
Arm/Group | PROPEL Mini Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 46 | 47
Number analyzed (Sinuses) | 46 | 47
mm | 43.2 (32.22) | 45.8 (36.29)
Statistical Analysis 1: Comparison: PROPEL Mini Sinus Implant vs Balloon Sinus Dilation Alone; Test type: Superiority; p = 0.68, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from enrollment through Day 180 post-procedure.
Description: Adverse event data were collected by clinical investigators using MedDRA terms, organized by System Organ Class.
Groups:
- All Participants: An intra-patient control design with placement of the Propel Mini Sinus Implant in one frontal sinus ostia (FSO) assigned to the treatment group following in-office balloon dilation compared to in-office balloon dilation without implant placement of the contralateral frontal sinus ostia (FSO) assigned to the control group.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 5/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=50)
Acute sinusitis (Infections and infestations) | 3 (3)
Vision blurred (Nervous system disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
One limitation of this study design is utilizing an intra-patient control. This precludes evaluation of patient-reported outcomes. However, it also minimizes interpatient variability, and the differences in surgical techniques.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No